CLINICAL TRIAL: NCT03944070
Title: Management of Patients With Neovascular Age-related Macular Degeneration Undergoing Cataract Surgery: A Pilot Study
Brief Title: Management of Patients With Neovascular Age-related Macular Degeneration Undergoing Cataract Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ophthalmica Eye Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/001_OPH-ECSAMD
Record Dates: First submitted 2019-04-23; First posted 2019-05-09 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Wet Macular Degeneration; Cataract Extraction
MeSH Terms: conditions — Wet Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Treatment (Active Comparator): The participants will receive x1 intraoperative and 3 postop monthly injections. Subsequently, they will follow the treat and extend protocol.
  Interventions: Drug: Ranibizumab
- Standard Treatment (Active Comparator): The participants will continue their preoperative treat and extend protocol .
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Intravitreal Ranibizumab is approved for the treatment of wet AMD. In this study we will compare an intensive injection protocol versus the standard treat and extend protocol in wet AMD patients undergoing cataract surgery.
  Other Names: Lucentis

SUMMARY:
To-date there have been only very few studies to examine the effect of cataract surgery to patients with wet age-related macular degeneration. The evidence on the effects of cataract surgery in such patients suggests improvement of their visual function and quality of life, but at the same time a subclinical susceptibility to macular edema and exacerbation of the choroidal neovascularization. Therefore it is highly important to identify the optimum treatment regime, pursuing the best anatomical and functional postoperative results.

DETAILED DESCRIPTION:
To-date there have been only very few studies to examine the effect of cataract surgery to patients with neovascular age-related macular degeneration (AMD), especially in the era of anti-vascular endothelial growth factor (anti-VEGF) therapy. Furthermore the issue of optimum treatment regimen that should be used in the peroperative period has never been addressed. Since the human life expectancy gradually increases, the number of patients who are under anti-VEGF intravitreal injections for wet AMD will be increasing accordingly. Cataract surgery in such patients, despite guarded prognosis has been proved to improve their visual function and quality of life. On the other hand, it has been shown that cataract surgery induces anatomic changes based on optical coherence tomography analysis, suggesting a subclinical susceptibility to postoperative cystoid macular edema or exacerbation of choroidal neovascularization. Therefore it is highly important to identify the optimum treatment regime, pursuing the best anatomical and functional postoperative results.

ELIGIBILITY:
Inclusion Criteria:

* Active choroidal neovascularization (at least 1 intravitreal injection in the past 12 months) associated with AMD and involving the foveal center
* BCVA of 1.0 (LogMAR) or better
* Duration of wet AMD less than 3 years

Exclusion Criteria:

* Coexisting ocular pathology potentially affecting visual acuity and/or status of the macula including diabetic retinopathy, advanced glaucoma, retinal vein occlusion, retinal detachment
* Newly diagnosed patients with wet AMD who are on anti-VEGF treatment for less than 6 months

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Visual acuity change from baseline | 12 months
  Difference in visual acuity change from baseline at the end of the follow-up period.
Difference in the number of injections | 12 months
  Difference in the number of injections at the end of the follow-up period.

SECONDARY OUTCOMES:
Status of the macular degeneration based on optical coherence tomography parameter, as compared to baseline | 12 months
  The status of the age-related macular degeneration will be evaluated based on optical coherence tomography parameters at the at final follow-up and compared to the baseline. Our main focus is to identify any subfoveal scarring and/ or subfoveal atrophy that may develop during the follow-up and assess changes from the baseline state of the macula.

CONTACTS AND LOCATIONS:
Overall Officials: Paris G Tranos, PhD, Principal Investigator — Head of Uveitis & Retinal Surgery Department, Ophthalmica Eye Institute
Locations (1):
- Ophthalmica Eye Institute, Thessaloniki, Kalamaria, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kessel L, Erngaard D, Flesner P, Andresen J, Tendal B, Hjortdal J. Cataract surgery and age-related macular degeneration. An evidence-based update. Acta Ophthalmol. 2015 Nov;93(7):593-600. doi: 10.1111/aos.12665. Epub 2015 Jan 20. PMID 25601333
- [Background] Saraf SS, Ryu CL, Ober MD. The effects of cataract surgery on patients with wet macular degeneration. Am J Ophthalmol. 2015 Sep;160(3):487-492.e1. doi: 10.1016/j.ajo.2015.06.006. Epub 2015 Jun 19. PMID 26095263